CLINICAL TRIAL: NCT01877343
Title: Developing a Non-invasive Cardiac Functional Health Status Measurement Device to be Used in a Critical Population of Adults and Children With Heart Failure.
Brief Title: Developing a Non-invasive Cardiac Functional Health Status Measurement Device
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Challenges associated with study enrollment due to stress test, study terminated
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB201300055
Record Dates: First submitted 2013-04-15; First posted 2013-06-13 (Estimated); Results first posted 2016-02-10 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Heart Failure
Keywords: cardiac functional health classification; Congenital heart failure; chronic heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CVInsight (TM) (Experimental): Patient will be placed on a tilt table and pulse oximetry (Nonin Medical)and blood pressure will be measured at different table positions (different angles). A hemodynamic monitor called CVInsight(TM) will be used to monitor the pulse oximeter readings.
  Interventions: Device: CVInsight(TM)

INTERVENTIONS:
Device: CVInsight(TM) — Patient will be placed on a tilt table and pulse oximetry (Nonin Medical) and blood pressure will be measured at different table positions (different angles). Four positions will be explored. A hemodynamic monitor called CVInsight(TM) will be used to monitor the pulse oximeter readings.

SUMMARY:
This is a single-center, non-randomized study.Enrolled patients will be placed on a tilt table and a stress test will be performed in a total of 4 different positions. Their blood pressure will be measured at each position. Also, a pulse oximeter will be placed on the forehead to measure pulse rate and strength. These results will be compared to cardiac functional classifications defined by New York Heart Association (NYHA) criteria for adults and New York Pediatric Heart Failure (NYPHF) index for our pediatric age patients. The primary aim of this initiative is to assess the discriminatory value of a cardiac functional health classification based upon the degree of dependency of cardiac function on changes in cardiac preload and afterload circulatory volume.

DETAILED DESCRIPTION:
Participants will be asked to review the informed consent and consent to the study prior to any study procedures. The study will consist of a single visit to the Medical Plaza at the University of Florida. During this visit, Enrolled patients will be placed on a tilt table and their position changed to a total of 4 different positions. Their blood pressure will be measured at each position. Also, a pulse oximeter will be placed on the forehead to measure pulse rate and strength. The study will take approximately 25 minutes. Data collected shall include a questionnaire for the patient, a list of the patient's co-morbidities, an echocardiogram or catheter lab data if available, and a list of the patient's current medications.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure patient eligibility shall consist of the following:

Group 1a: 5 adult heart transplant patients

* Age ≥ 21 years old and <74 years old
* Speaks and understands English
* Provides Informed Consent

Group 1b: 5 pediatric heart transplant patients

* Age ≥ 7 years old and < 21 years old
* Speaks and understands English
* Provides Informed Consent

Group 2: 5 adult heart failure patients

* Age ≥ 21 years old and <74 years old
* Speaks and understands English
* Provides Informed Consent

Group 3: 5 adult aged Fontan patients

* Age ≥ 21 years old and <74 years old
* Speaks and understands English
* Provides Informed Consent

Group 4: 5 pediatric Fontan patients

* Age ≥ 7 years old and < 21 years old
* Speaks and understands English
* Provides Informed Consent

Group 5: 5 pediatric patients limited to heart murmurs

* Age ≥ 7 years old and < 21 years old
* Speaks and understands English
* Provides Informed Consent

Group 6: 5 normal adult patients

* Age ≥ 21 years old and <74 years old
* Speaks and understands English
* Provides Informed Consent

Exclusion Criteria:

* • Unstable patients per judgment of the clinician prior to the start of the treatment

  * Patients unable to have blood pressure cuff measured on the upper arm
  * Inability to wear monitor on forehead
  * Patients will be excluded from the study if they have eaten, consume caffeinated beverages, or taken hypertensive medications within 2 hours of testing

Ages: 7 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Curt DeGroff, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients recruited only from two of the study groups (control and post-transplant). Patients from the other groups were not included as study team assessed feasibility with the non-heart failure groups prior to consenting high failure patients. Enrollment was challenging for high risk patients due to stress test severity.
Groups:
- Adult Heart Transplant (1a); Pediatric Heart Tansplant (1b); Adult Heart Failure; Adult Fontan; Pediatric Fontan; Pediatric Controls; Adult Controls: Patient will be placed on a tilt table and pulse oximetry (Nonin Medical)and blood pressure will be measured at different table positions (different angles). A hemodynamic monitor called CVInsight(TM) will be used to monitor the pulse oximeter readings.
  CVInsight(TM): Patient will be placed on a tilt table and pulse oximetry (Nonin Medical) and blood pressure will be measured at different table positions (different angles). Four positions will be explored. A hemodynamic monitor called CVInsight(TM) will be used to monitor the pulse oximeter readings.
Period: Overall Study
Arm/Group | Adult Heart Transplant (1a) | Pediatric Heart Tansplant (1b) | Adult Heart Failure | Adult Fontan | Pediatric Fontan | Pediatric Controls | Adult Controls
Started | 2 | 3 | 0 | 0 | 0 | 5 | 0
Completed | 2 | 3 | 0 | 0 | 0 | 5 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pediatric Heart Transplant (1b); Pediatric Controls: Patient will be placed on a tilt table and pulse oximetry (Nonin Medical)and blood pressure will be measured at different table positions (different angles). A hemodynamic monitor called CVInsight(TM) will be used to monitor the pulse oximeter readings.
  CVInsight(TM): Patient will be placed on a tilt table and pulse oximetry (Nonin Medical) and blood pressure will be measured at different table positions (different angles). Four positions will be explored. A hemodynamic monitor called CVInsight(TM) will be used to monitor the pulse oximeter readings.
- Total: Total of all reporting groups
Arm/Group | Adult Heart Transplant (1a) | Pediatric Heart Transplant (1b) | Pediatric Controls | Total
Number analyzed (Participants) | 2 | 3 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 2 | 5 | 7
  Between 18 and 65 years | 2 | 1 | 0 | 3
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 7
  Male | 0 | 1 | 2 | 3
Height [Mean (Standard Deviation); unit: meters] | 1.736 (.004) | 1.62 (.03) | 1.64 (.1) | 1.65 (.09)
Weight [Mean (Standard Deviation); unit: kg] | 83 (15) | 77 (25) | 56 (11) | 67 (21)
BMI [Mean (Standard Deviation); unit: kg/m2] | 27.4 (5.0) | 28.9 (8.7) | 20.5 (1.7) | 24.4 (6.7)

OUTCOME MEASURES:

1. Primary Outcome: Pulse Rate
Description: Continuous change of pulse rate from baseline through the end of the study will be followed. Changes in pulse rate will be plotted against the four tilt table positions. Four positions will be explored, Mounting position, baseline, passive leg raise (cardiac preload dependent) and orthostasis head raise (cardiac afterload dependent). Patients go from mounting position, to baseline, to the corresponding position (passive leg raise or orthostasis head raise) and back to baseline. The assessment will take 30 minutes. From the graph, average pulse rate is calculated.
Time Frame: Average pulse rate from baseline to 30 minutes
Population: The study was terminated and the data was not sent to the contract company to analyze. The software package to compile the data is not available to the University of Florida.
Arm/Group | CVInsight (TM)
Number analyzed (Participants) | 0

2. Primary Outcome: Pulse Strength
Description: Continuous change of pulse strength from baseline through the end of the study. Pulse strength is measured as volts by the system. Changes in pulse strength will be plotted against the four tilt table positions. Four positions will be explored, Mounting position, baseline, passive leg raise (cardiac preload dependent) and orthostasis head raise (cardiac afterload dependent). Patients go from mounting position, to baseline, to the corresponding position (passive leg raise or orthostasis head raise) and back to baseline. The assessment will take 30 minutes. Cardiac function curves will be constructed with the data collected and average pulse strength from baseline to 30 minutes will be reported.
Time Frame: Average pulse strength from baseline to 30 minutes
Population: as for outcome 1
Arm/Group | CVInsight (TM)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | CVInsight (TM)
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
Early termination due concerns for severity of stress test on high risk patients. Only control and post-transplant groups had enrollment. Statistical analysis cannot be performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes